CLINICAL TRIAL: NCT06093386
Title: Promoting Intensive Transitions for Children and Youth With Medical Complexity From Pediatric to Adult Care
Acronym: PITCare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Eyal Cohen, Program Head and Senior Scientist, Child Health Evaluative Sciences, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1000080621
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Children and Youth With Medical Complexity
Keywords: transition; complex care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Intensive Transition Support
- Control/ Usual Care (No Intervention): Standard of care in the control group will involve the utilization of existing tools within clinical programs which may include preparation for transitions, but there will be no systematic follow-up by a paediatric provider beyond age 18. Care will be transferred to adult providers (primary care and specialists) via a transition guide that will be offered to participants and their referring providers. This is the current model of care for virtually all CMC in Ontario.

INTERVENTIONS:
Other: Intensive Transition Support — Participants assigned to the intervention arm will transfer their transition support leadership to a transition team composed of a transition navigator (an advance practice nurse), a nurse navigator (a registered nurse) and a social worker over 2 years to support them through the multiple phases of CMC transitions including guidance, monitoring, planning, care transfer and transfer completion. CMC and their caregivers will be offered support in care planning, receiving funding, and connecting with a primary care provider and adult subspecialists.
  Arms: Intervention

SUMMARY:
Medical advances have allowed many more children and youth with medical complexity (CMC) to survive well into adulthood. However, this has not been matched with increases in knowledge of complex conditions or the availability of supports as they transition into the adult care system. The goal of this randomized control trial is to compare intensive transition support from a transition team, led by an advance practice nurse, during transition to adult care for 2 years, with usual care in CMC. Participants assigned to the intervention group will be offered support in care planning, receiving funding, and connecting with a primary care provider and adult subspecialists.

The main questions it aims to answer are:

1. Does intensive transition support improve the patient's continuity of care over 2 years compared with usual care?
2. Will there be differences between intervention and control groups with respect to other outcomes related to the youth/family's satisfaction with care, care coordination, self-care, health service utilization, cost-effectiveness, and quality of life?
3. What are the experiences of youth, parents, the transition team, and other clinicians involved in the intensive transition support process?

ELIGIBILITY:
Inclusion Criteria:

* Patients 17 years 6 months- 17 years 9 months old (inclusive) who meet Ontario's CMC definition:

  1. technology dependence and/or users of high-intensity care,
  2. fragility (severe and/or life-threatening condition,
  3. chronicity (expected to last at least 6 months),
  4. complexity (involvement of ≥5 healthcare practitioners/teams and healthcare services in ≥ 3 locations such as home, school, hospital, etc.).

Exclusion Criteria:

* are expected to die within 2 years of recruitment (e.g., those receiving active end-of-life care)
* do not have a stable primary caregiver (e.g., those who reside in residential or long-term care facilities, and those in foster care as the intervention is focused on a patient-caregiver dyad)

Ages: 210 Months to 213 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Transfer Completion | 6 to 30 months
  Successful transfer of primary and subspecialty care to continuous primary care and a prioritized subspecialty in adult care will be measured using a relational continuity of care measure - the Bice Boxerman Index (modified for the study population).

SECONDARY OUTCOMES:
Transfer Completion | Baseline to 24 months
  Successful transfer of primary and subspecialty care to continuous primary care and a prioritized subspecialty in adult care will be measured using a relational continuity of care measure - the Bice Boxerman Index (modified for the study population).
Transfer Completion | 6 to 30 months
  Successful transfer of primary care to continuous adult primary care will be measured using a relational continuity of care measure - the Bice Boxerman Index.
Transfer Completion | 6 to 30 months
  Successful transfer of subspecialty care to continuous care from a prioritized subspeciality provider in adult care will be measured using a relational continuity of care measure - the Bice Boxerman Index.
Transfer Completion | Baseline to 24 months
  Successful transfer of subspecialty care to continuous care from all subspecialty providers in adult care will be measured using a relational continuity of care measure - the Bice Boxerman Index.
Transfer Completion | Baseline to 24 months
  The proportion of patients who receive a Bice Boxerman Index score of 0 (< 2 visits to both a subspecialty and primary care provider) will be assessed.
Transfer Completion | Baseline to 24 months
  The proportion of visits to all primary care providers that are made to the usual care provider will be assessed among individuals who had ≥ 3 primary care visits (UPC Index).
Early Identification and Transition Readiness- Satisfaction with Transitional Healthcare | Baseline, 12 months and 24 months
  The change in caregiver satisfaction with transitional health care services will be measured using the Larsen Client Satisfaction Questionnaire (CSQ) (8-item). The change in patient satisfaction will also be measured with the CSQ where able. Comparisons will be made between intervention and control groups.
Early Identification and Transition Readiness- Self-Care | Baseline, 12 months and 24 months
  The change in the caregiver's family empowerment status will be measured with the Family Empowerment Scale (24-item). Scoring will be accomplished by summing responses from items within the family (12 items) and service system (12 items) to generate sub-scores. Comparisons will be made between intervention and control groups.
Early Identification and Transition Readiness- Self-Care | Baseline
  The change in the patient's knowledge and confidence in managing their health will be measured (if able) using the Patient Activation Measure (10-item). Comparisons will be made between intervention and control groups.
Information Sharing and Support, Transition Plan and Coordinated Transition | Baseline, 12 months and 24 months
  The change in utility of care planning tools, written transition plan assessment, coordination of care among providers and families and, coordination of care between providers and families will be assessed with the Family Experiences with Coordination of Care (FECC) survey, completed by the caregiver. Comparisons will be made between intervention and control groups.
Introduction to Adult Services | 24 months
  The number of patients who have received (presence or absence) adult-oriented funding and services will be assessed via report by the caregiver or, if able, the youth (e.g., receipt of Ontario Disability Support Program ODSP funding). Comparisons will be made between intervention and control groups.
Use of Services | Baseline to 24 months
  Low acuity emergency department visits, emergency department use, hospitalization, technological complications, and immunization will be captured using encoded health administrative data housed at ICES to determine the patient's health care and preventative care use. Comparisons will be made between intervention and control groups.
Use of Services- Incremental Cost-Utility Ratio (ICUR) | Baseline to 24 months
  A probabilistic cost-utility analysis will be conducted using patient-level data, to determine the incremental cost per quality-adjusted life-year gained (QALY) of intensive transition support compared to usual care, from a health system perspective. QALY gains for both patient and caregiver will be included. All direct health care costs and health service utilization will be ascertained from study data linked to administrative datasets at ICES. Utility, determined by mapping patient and caregiver responses to the EQ-5D-5L, will be used to generate QALY gains (or losses) over the time horizon.
Health-Related Quality of Life | Baseline, 12 months and 24 months
  The change in overall health-related quality of life of both the patient and their caregiver will be measured using the EQ-5D-5L. The digit for each of the scale's five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) can be combined into a 5-digit number that describes the patient's health state and is commonly used to estimate health utilities. The descriptive system is complemented by a visual analogue scale where patients record their self-rated health. Comparisons will be made between intervention and control groups.
Health-Related Quality of Life-Caregiver Fatigue | Baseline, 12 months and 24 months
  The change in caregiver fatigue will be measured using the PROMIS Fatigue Scale (8-item). The Fatigue scale is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. Each question has five response options ranging in value from one to five. Comparisons will be made between intervention and control groups.
Health-Related Quality of Life- Family Distress | Baseline, 12 months and 24 months
  The change in family distress will be assessed using the Brief Family Distress Scale (1-item) completed by the caregiver. The 10-point Likert scale is used to measure crisis level, which is assigned by groupings of the scale continuum, with a level between 1-3 indicating no impairment, 4-5, moderate impairment, and 6-10, marked impairment. Comparisons will be made between intervention and control groups.
Experiences in The Process | 12 to 24 months
  Semi-structured qualitative interviews will be conducted with a subset of intervention participants, health care providers, including both pre-transition and post-transition clinicians, and the transition team to gauge their experience with the transition support process.

OTHER OUTCOMES:
Implementation Progress Outcomes- Care Planning | Baseline to 24 months
  The implementation process will be assessed by determining the fidelity of the intervention using percentages of completion for each of the four main intervention components. The percentage of completed care planning documentation will be captured by the transition team for those participants assigned to the intervention group.
Implementation Progress Outcomes- Integration with Primary Care Providers | Baseline to 24 months
  The implementation process will be assessed by determining the fidelity of the intervention using percentages of completion for each of the four main intervention components. The percentage of primary care visits scheduled and attended by the transition team will be captured by the transition team for those participants assigned to the intervention group.
Implementation Progress Outcomes- Adult Subspecialty Facilitation | Baseline to 24 months
  The implementation process will be assessed by determining the fidelity of the intervention using percentages of completion for each of the four main intervention components. The percentage of joint adult subspecialty visits and visits scheduled and attended by the transition team will be captured by the transition team for those participants assigned to the intervention group.
Implementation Progress Outcomes- Facilitation of Funding | Baseline to 24 months
  The implementation process will be assessed by determining the fidelity of the intervention using percentages of completion for each of the four main intervention components. The percentage of eligible funding applications completed and received will be captured by the transition team for those participants assigned to the intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santos S, Thomson D, Diaz S, Soscia J, Adams S, Amin R, Bernstein S, Blais B, Bruno N, Colapinto K, Espin S, Fayed N, Greenaway J, Henze M, Ivers NM, LeGrow K, Lim A, Lippett R, Lunsky Y, Macarthur C, Mahant S, Malecki S, Miranda S, Moharir M, Moretti ME, Phillips L, Robeson P, Taryan M, Thorpe K, Toulany A, Vandepoele E, Weitzner B, Orkin J, Cohen E. Promoting Intensive Transitions for Children and Youth with Medical Complexity from Paediatric to Adult Care: the PITCare study-protocol for a randomised controlled trial. BMJ Open. 2024 Dec 9;14(12):e086088. doi: 10.1136/bmjopen-2024-086088. PMID 39653557